CLINICAL TRIAL: NCT03863613
Title: The Effectiveness of Cervical Pessary Compared to Cervical Cerclage With or Without Vaginal Progesterone for the Prevention of Preterm Birth in Women With a Twin Pregnancy and a Short Cervix: a Two-by-two Factorial Randomised Clinical Trial
Brief Title: Pessary Versus Cerclage With or Without Progesterone in Twins
Acronym: PCP-Twins
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to safety concerns as the PTB <28 weeks and perinatal death rates were significantly higher in the pessary group, following the DSMC's recommendation.
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CS/MD/19/01
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-12

CONDITIONS: Preterm Birth; Twin Pregnancy; Short Cervix
Keywords: Pessary, Cerclage, Progesterone, Twins, Preterm birth
MeSH Terms: conditions — Premature Birth | interventions — Pessaries; Cerclage, Cervical; Progesterone

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to either cerclage, pessary, cerclage plus progesterone or pessary plus progesterone in a 1:1:1:1 ratio with a variable block size of 4 or 8.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pessary group (Active Comparator): A soft, flexible, silicone pessary, purchased from the manufacturer (Arabin®, Dr Arabin GmbH & Co KG, Germany) will be inserted through the vagina, upward around the cervix by 4 senior clinicians, who had experienced with pessary used, within one week of randomisation. Size of the pessary will be determined at the time of speculum inspection.
  Interventions: Device: Pessary
- Cerclage group (Active Comparator): Women will be receiving the cervical cerclage according to local protocol, within a week after randomisation. 3 senior clinicians who had experienced with cerclage, will perform cerclage, using Mc Donald technique, under spinal anaesthesia.
  Interventions: Procedure: Cervical cerclage
- Pessary plus progesterone group (Active Comparator): 400 mg vaginal progesterone, purchased from the manufacturer (Cyclogest® 400mg, Actavis, United Kingdom), will be applied once daily at bedtime, starting from the day of randomisation, in addition to the pessary that has been placed. Participants will be asked to record their drug application in a patient diary sheet for up to 140 days.
  Interventions: Device: Pessary; Drug: Vaginal progesterone
- Cerclage plus progesterone group (Active Comparator): 400 mg vaginal progesterone, purchased from the manufacturer (Cyclogest® 400mg, Actavis, United Kingdom), will be applied once daily at bedtime, starting from the day of randomisation, in addition to the cerclage that has been placed. Participants will be asked to record their drug application in a patient diary sheet for up to 140 days.
  Interventions: Procedure: Cervical cerclage; Drug: Vaginal progesterone

INTERVENTIONS:
Device: Pessary — A soft, flexible, silicone pessary (Arabin®, Dr Arabin GmbH & Co KG, Germany) will be inserted through the vagina, upward around the cervix.
  Other Names: Arabin
  Arms: Pessary group; Pessary plus progesterone group
Procedure: Cervical cerclage — Cervical cerclage using Mc Donald technique, under anaesthesia
  Other Names: Stitch
  Arms: Cerclage group; Cerclage plus progesterone group
Drug: Vaginal progesterone — Cyclogest® 400mg, Actavis, United Kingdom, applied once daily at bedtime
  Other Names: Cyclogest 200 mg
  Arms: Cerclage plus progesterone group; Pessary plus progesterone group

SUMMARY:
This study compares the effectiveness of cervical pessary and cervical cerclage with or without vaginal progesterone for prevention of preterm birth in women with a twin pregnancy and a cervix ≤28 mm.

Participants will be randomly assigned in a 1:1:1:1 ratio to receive cerclage, pessary, cerclage plus progesterone or pessary plus progesterone.

DETAILED DESCRIPTION:
This open label, multi-center, two-by-two factorial, randomised controlled trial aims to compare the effectiveness of cervical pessary to cervical cerclage and also to determine the effectiveness of vaginal progesterone for the prevention of PTB in women with a twin pregnancy and a cervix ≤28 mm.

All women with a twin pregnancy will undergo cervical length measurement and digital examination at screening. Prior to CL measurement, women will be given a short brochure outlining risk factors and available PTB prevention methods. Only women with a CL ≤28 mm will be eligible for the study. Eligible participants will be screened by midwives or gynaecologists, then participants will be provided a full participant Information Sheet, Consent Form and will be invited to a full discussion with investigators about the study. Eligible women will further undergo a speculum examination to assess the feasibility of treatment with either cerclage or cervical pessary with or without progesterone and to exclude premature rupture of the membranes (PROM), acute vaginitis and cervicitis. All eligible women will be invited to participate in the study.

After written informed consent, women will be randomly assigned in a 1:1:1:1 ratio to receive a cerclage, pessary, cerclage plus progesterone or pessary plus progesterone. Assignment to treatment allocation will be done via a web portal hosted by HOPE Research Center, Vietnam. The randomisation schedule will be computer-generated at HOPE Research Center, with a permuted random block size of 4 or 8. Blinding will not be possible due to the nature of interventions. However, neonatologists assessing the children will be unaware of treatment allocation. Apart from randomisation, patients will be followed up and treated according to local protocol.

Women allocated to a cervical cerclage will be receiving the intervention according to local protocol, within a week after randomisation. Briefly, 2 to 3 senior clinicians, who had experienced with cerclage, will perform cervical cerclage, using Mc Donald technique, under spinal anaesthesia with a single dose of prophylactic antibiotics.

For those who randomised to pessary group, a soft, flexible, silicone pessary, purchased from the manufacturer (Arabin®, Dr Arabin GmbH & Co KG, Germany), will be inserted through the vagina, upward around the cervix by 4 senior clinicians, who had experienced with pessary used, within one week of randomisation. The size of the pessary will be determined at the time of speculum inspection (Arabin and Alfirevic, 2013).

In the cerclage plus progesterone group, 400 mg vaginal progesterone, purchased from the manufacturer (Cyclogest® 400mg, Actavis, United Kingdom), will be applied once daily at bedtime, within two days after cerclage insertion. Participants will be asked to record their drug application in a patient diary sheet for up to 140 days.

In the pessary plus progesterone group, 400 mg vaginal progesterone, purchased from the manufacturer (Cyclogest® 400mg, Actavis, United Kingdom), will be applied once daily at bedtime, within two days after pessary insertion, in addition to the pessary that has been placed. Participants will be asked to record their drug application in a patient diary sheet for up to 147 days.

In all groups, participants will be re-assessed at 14 days post-randomisation for any possible adverse event. After that, participants will be seen monthly or weekly per local protocol. CL measurement will not be performed routinely after randomisation, unless for patients' preference. In case the CL was shortened, further intervention, if any, will be based on the clinician's decision after a discussion with the patient.

In case of premature rupture of the membranes, active vaginal bleeding, other signs of preterm labor or severe patient discomfort, the vaginal progesterone and pessary or cerclage, will be removed. If participants develop (threatened) preterm labor, participants will receive treatment per local protocol. Intervention will be stopped at 37 0/7 weeks of gestation or at delivery.

Compliance rate to progesterone will be calculated by dividing the number of progesterone doses used since the last visit by the number of progesterone doses that should have been used since the last visit. Women will be defined as compliant when the compliance rate are over 80%.

Statistical analysis will be conducted according to the intention-to-treat principle, in which all randomised women will be considered in the primary comparison between treatment groups. The per-protocol analysis may be conducted, but these results would be considered exploratory only. All tests will be two-tailed, and differences with p-value <0.05 will be considered statistically significant.

In view of the two-by-two factorial design, the analysis will be done separately for cerclage versus pessary and for progesterone versus no progesterone. The investigators will test for interaction between CL and treatment effect on PTB <34 weeks and the composite of poor perinatal outcomes.

A pre-specified subgroup analysis in women with a CL <25th percentile, and at the 25-50th percentile, 50-75th percentile and >75th percentile is planned. The percentile will be determined based on the CL from all women after randomisation.

The investigators plan one interim analysis. The interim analysis will be performed by an independent statistician who will not directly involve in the study, after completion of data collection of the first 150 randomised patients. At interim analyses, data will be assessed for safety, efficacy, and futility. Safety will be assessed in terms of serious adverse events (perinatal death, maternal mortality or severe maternal morbidity). The interim analysis will be conducted using a two-sided significant test with the Haybittle-Peto spending function and a type I error rate of 5% with stopping criteria of p <0.001 (Z alpha = 3.29). Based on this report, the DSMB will provide guidance on whether to stop or continue the study.

A separated detailed statistical analysis plan will be developed and completed prior to data lock.

Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) and study protocol will be available, upon request from investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose to achieve aims in the approved proposal. Data will be available at the beginning 9 months and ending 36 months following article publication. Proposals should be directed to bsvinh.dq@myduchospital.vn. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at https://www.project-redcap.org/.

ELIGIBILITY:
Inclusion Criteria:

* Women with a twin pregnancy (mono- and di-chorionic)
* 16 0/7 to 22 0/7 weeks of gestation
* Maternal age ≥18 yrs
* Cervical length ≤28 mm
* Informed consent
* Not participating in another preterm birth study at the same time

Exclusion Criteria:

* Uterine anomalies
* Cervical dilation with visible amniotic membranes or amniotic membranes prolapsed into the vagina
* Twin-to-twin transfusion syndrome
* Stillbirth or major congenital abnormalities in any of the fetus
* Severe vaginal discharge
* Acute vaginitis or cervicitis
* Vaginal bleeding
* Placental preavia
* Vasa preavia
* Premature rupture of membranes
* Premature labor with/without ruptured membrane
* Suspicion of chorioamnionitis
* Cerclage or pessary in place or unable to undergo cervical cerclage or pessary

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Preterm birth <34 weeks | From date of randomisation until 33 6/7 weeks
  Birth before 34 weeks' gestation

SECONDARY OUTCOMES:
Gestational age at delivery | At birth
  Gestational age at delivery Time from randomisation to delivery Delivery < 24 weeks, < 28 weeks, < 32 weeks and < 37 weeks of gestation Spontaneous preterm birth < 24 weeks, < 28 weeks, < 32 weeks and < 37 weeks of gestation Onset of labor: spontaneous, labor induction, elective C-section Mode of delivery: vaginal delivery, C-section All livebirths at any gestational age Use of tocolytic drugs Use of antenatal corticosteroids Use of magnesium sulfat for fetal neuroprotection Preterm prelabour rupture of membranes Length of maternal admission for preterm labor (days) Chorioamnionitis Marternal mortality
Time from randomisation to delivery | From date of randomisation until the date of delivery, assessed up to 22 weeks
  Time interval between randomisation and delivery
Preterm birth <28 weeks | From date of randomisation until 27 6/7 weeks
  Birth before 28 weeks' gestation
Preterm birth <37 weeks | From date of randomisation until 36 6/7 weeks
  Birth before 37 weeks' gestation
Spontaneous preterm birth <28 weeks | From date of randomisation until 27 6/7 weeks
  Birth spontaneously before 28 weeks' gestation, including preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM)
Spontaneous preterm birth <34 weeks | From date of randomisation until 33 6/7 weeks
  Birth spontaneously before 34 weeks' gestation, including preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM)
Spontaneous preterm birth <37 weeks | From date of randomisation until 36 6/7 weeks
  Birth spontaneously before 37 weeks' gestation, including preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM)
Iatrogenic preterm birth <28 weeks | From date of randomisation until 27 6/7 weeks
  Birth non-spontaneously before 28 weeks' gestation
Iatrogenic preterm birth <34 weeks | From date of randomisation until 33 6/7 weeks
  Birth non-spontaneously before 34 weeks' gestation
Iatrogenic preterm birth <37 weeks | From date of randomisation until 36 6/7 weeks
  Birth non-spontaneously before 37 weeks' gestation
Onset of labor | At birth
  Spontaneous, labor induction, elective C-section
Mode of delivery | At birth
  Vaginal delivery, C-section (elective, suspected fetal distress, non-progressive labor)
Livebirth | At birth
  The birth of at least one newborn, regardless of gestational age, that exhibits any sign of life such as respiration, heartbeat, umbilical pulsation or movement of voluntary muscles
Use of tocolytic drugs | From 24 0/7 to 33 6/7 weeks' gestation
  Use of any tocolytic drug to treat preterm labour
Use of antenatal corticosteroids | From 24 0/7 to 33 6/7 weeks' gestation
  Use of antenatal corticosteroids to prevent respiratory distressed syndrome
Use of MgSO4 for neuroprotection | From 28 0/7 to 31 6/7 weeks' gestation
  Use of MgSO4 for neuroprotection in
Preterm prelabour rupture of membranes | From randomization to less than 37 weeks, up to 21 weeks
  Prelabour rupture of membranes and gestational age less than 37 weeks
Length of maternal admission for preterm labour | From 24 weeks to 37 week
  Number of admission days for treatment of preterm labour
Chorioamnionitis | From randomization to delivery, up to 22 weeks
  Intraamniotic infection
Maternal mortality | From randomization to delivery, up to 22 weeks
  Death of the mother
Birthweight | At birth
  Weight of baby born
Birthweight <1500 g | At birth
  Weight of baby born <1500g
Birthweight <2500 g | At birth
  Weight of baby born <2500g
Congenital anomalies after randomisation | At birth
  Any congenital anomalies detected in baby born
5-min Apgar score | At birth
  Apgar score at 5 minute after birth
5-min Apgar score <7 | At birth
  Apgar score at 5 minute after birth <7
Admission to neonatal intensive care unit (NICU) | Within 7 days after birth
  Admission to neonatal intensive care unit of baby
Length of NICU admission | Up to 28 days after birth
  Number of admission days to NICU
Respiratory distress syndrome | Up to 28 days after birth
  The presence of tachypnoea >60/minute, sternal recession and expiratory grunting, need for supplemental oxygen, and a radiological picture of diffuse reticulogranular shadowing with an air bronchogram
Periventricular haemorrhage II B or worse | Up to 28 days after birth
  Repeated neonatal cranial ultrasound by the neonatologist according to the guidelines on neuro-imaging described by de Vries et al
Necrotizing enterocolitis | Up to 28 days after birth
  Diagnosed according to Bell
Proven sepsis | Up to 28 days after birth
  The combination of clinical signs and positive blood cultures
Stillbirth | At birth
  Baby born with no signs of life at or after 28 weeks' gestation
Death before discharge | Up to 28 days after birth
  Death of newborn before discharge from nursery
Composite of poor perinatal outcomes | Up to 28 days after birth
  Foetal or neonatal death, intraventricular haemorrhage, respiratory distress syndrome, necrotizing enterocolitis or neonatal sepsis
Maternal side effects | From date of randomisation until delivery, which is up to 22 weeks
  Including vaginal discharge, fever, vaginal bleeding, vaginal infection (confirmed by vaginal discharge culture), vaginal pain, pessary repositioning and necrosis or rupture of the cervix
Fetal death <24 weeks | From randomization to 23 6/7 weeks
  Fetal death before 24 weeks' gestation

CONTACTS AND LOCATIONS:
Overall Officials: Yen TN He, MD, Principal Investigator — My Duc Phu Nhuan Hospital
Locations (1):
- My Duc Phu Nhuan Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) and study protocol will be available, upon request from investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose to achieve aims in the approved proposal. Data will be available at the beginning 9 months and ending 36 months following article publication. Proposals should be directed to bsvinh.dq@myduchospital.vn. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at https://www.project-redcap.org/
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Data will be available at the beginning 9 months and ending 36 months following article publication.
Access Criteria: To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at https://www.project-redcap.org/.
URL: https://www.project-redcap.org/.

REFERENCES:
- [Derived] He YTN, Pham HNH, Nguyen TC, Bui TQ, Vuong NT, Nguyen DTN, Le TV, Li W, Le CH, Ho TM, Mol BW, Dang VQ, Vuong LN. Cervical cerclage versus cervical pessary with or without vaginal progesterone for preterm birth prevention in twin pregnancies and a short cervix: A two-by-two factorial randomised clinical trial. PLoS Med. 2025 Feb 21;22(2):e1004526. doi: 10.1371/journal.pmed.1004526. eCollection 2025 Feb. PMID 39982935
- [Derived] Dang VQ, He YT, Pham HN, Trieu TT, Bui TQ, Vuong NT, Nguyen LM, Nguyen DT, Le TV, Li W, Le CH, Mol BW, Vuong LN. Effectiveness of cervical pessary compared to cervical cerclage with or without vaginal progesterone for the prevention of preterm birth in women with twin pregnancies and a short cervix: study protocol for a two-by-two factorial randomised clinical trial. BMJ Open. 2020 Jun 16;10(6):e036587. doi: 10.1136/bmjopen-2019-036587. PMID 32554744